CLINICAL TRIAL: NCT05971992
Title: Effect of Intestinal Microbiota Modulation Induced by the Chicory Inulin-type β-fructans on Metabolic Parameters and Biomarkers of the Gut-skin Axis in Chronic Skin Inflammation
Brief Title: INulin-type Fructans-induced Gut Microbiota Modulation Impact on GUT-SKIN Axis Parameters in Psoriasis
Acronym: INGUTSKIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Polish Academy of Sciences (Other)
Collaborators: University of Warmia and Mazury (Other); Warsaw University of Life Sciences (Other)
Responsible Party: Principal Investigator, Urszula Krupa-Kozak, Principal Investigator, Polish Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2022/45/B/NZ9/03004
Record Dates: First submitted 2023-07-14; First posted 2023-08-02 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Psoriasis
Keywords: prebiotics; inulin-type fructans; chronic skin inflammation; inflammatory mediators and cytokines; intestinal barrier permeability; Psoriasis Area and Severity Index; dysbiosis; metabolic dysregulation; nutritional status; anthropometric indices; indirect respirometry; functional multi-sugars absorption test; quality of life; characteristics of gut microbiota; short-chain fatty acids; immunohistological skin analysis; gene expression; oxidative stress; volatile organic compounds
MeSH Terms: conditions — Psoriasis; Dysbiosis | interventions — maltodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Prebiotic (Experimental): Adult women and men (N = 35) with mild psoriasis (Psoriasis Area and Severity Index; PASI < 10) will receive 15g of prebiotic (chicory-derived inulin-type β-fructans) daily for 8 weeks
  Interventions: Dietary Supplement: Chicory-derived inulin-type β-fructans
- Placebo (Placebo Comparator): Adult women and men (N = 35) with mild psoriasis (Psoriasis Area and Severity Index; PASI < 10) will receive 15g of placebo (maltodextrin) daily for 8 weeks
  Interventions: Dietary Supplement: Maltodextrin
- Control (No Intervention): Healthy adult women and men (N = 30) will not receive any dietary intervention

INTERVENTIONS:
Dietary Supplement: Chicory-derived inulin-type β-fructans — This supplement will be portioned into moisture-impermeable sachets containing 7.5 grams of prebiotic. During the first two weeks, to avoid eventual side effects, PS participants will be advised to consume the contents of one sachet at breakfast only. Starting in week 3 until the end of the 8-weeks intervention the participants will consume the content of two sachets daily (at breakfast and at dinner) resulting in a total dose of 15 grams of prebiotic per day. Participants will be provided with a package of sachets in the amount required for the whole 8-weeks nutritional intervention. They will be instructed to dissolve the sachet content with water or juice and to drink it 15-20 minutes prior to their regular meal. The medium for suspending the supplement (water or juice) could be chosen by the participants and could be changed during the study.
  Other Names: Orafti®Synergy1 (Beneo, Tienen, Belgium)
  Arms: Prebiotic
Dietary Supplement: Maltodextrin — This supplement will be portioned into moisture-impermeable sachets containing 7.5 grams of maltodextrin. During the first two weeks, to avoid eventual side effects, PS participants will be advised to consume the contents of one sachet at breakfast only. Starting in week 3 until the end of the 8-week intervention the participants will consume the content of two sachets daily (at breakfast and at dinner) resulting in a total dose of 15 grams of placebo per day. Participants will be provided with a package of sachets in the amount required for the whole 8-weeks nutritional intervention. They will be instructed to dissolve the sachet content with water or juice and to drink it 15-20 minutes prior to their regular meal. The medium for suspending the supplement (water or juice) could be chosen by the participants and could be changed during the study.
  Arms: Placebo

SUMMARY:
There is increasing evidence of a strong, bidirectional correlation between the gut and the skin, that associates gastrointestinal health with skin homeostasis and allostasis. The dysregulation in the intestinal microbiome-host interplay is connected with the development of many chronic skin inflammations.

Plaque psoriasis is a chronic, immune-mediated non-communicable dermatitis affecting approximately 2-3% of the world's population, regardless of gender and age. In most cases (about 70-80%), the skin lesions are mild and do not require systemic treatment. Its etiology is not fully understood, but apart from the genetic predisposition, it is strongly associated with the "gut-skin axis". The rise of the local and systemic immune response in psoriasis is a consequence of systemic inflammation due to intestinal dysbiosis associated with increased intestinal permeability. Thus, gut microbiota modulation should become a research target due to its great potential to impact inflammation, including skin dermatitis, and its manifested consequences.

Diet is an underestimated element in psoriasis management, meanwhile, the dietary ingredients support skin health. Among them, prebiotics favorably alters the composition and activity of the intestinal microbes and alleviates inflammation in the intestines. It was hypothesized that restoring the balance of the gut microbiome and the proper functioning of the intestinal barrier in subjects with psoriasis will alleviate the inflammatory symptoms and skin lesions observed in this chronic dermatitis.

The goal of this clinical trial is to determine if a diet supplementation with prebiotic (chicory-derived inulin-type β-fructans; ITFs) vs. placebo (maltodextrin) will induce health-related benefits in a mild degree PS, and determine if the identified benefits are evoked by compositional and/or functional shifts of the intestinal bacterial communities. Healthy individuals will constitute a control group (C).

DETAILED DESCRIPTION:
The gut microbiota contributes to the health of the host. It enables the digestion of food, the proper functioning of the immune system, and protection against the invasion of pathogens. The gut microorganisms play a key role in maintaining the integrity of the intestinal epithelium. The epithelium serves as a selective barrier that, on the one hand, separates the immune cells of the intestinal mucosa from the microorganisms present in the lumen of the gut, and at the same time allows microbial metabolites to interact with the host cells and thus regulate the immune response. Dysbiosis of the intestinal microflora may result in damage to the intestinal integrity and, consequently, an increase in the permeability of the intestinal barrier. The translocation of bacterial antigens and metabolites into the bloodstream contributes to the activation of the local and systemic immune response resulting in local and systemic inflammation. Disruption of the interaction between the gut microbiome and the host can lead to inflammation. Plaque psoriasis is a chronic, immune-mediated dermatitis. It is manifested by peeling, itching, and reddening of the skin. Psoriasis is a non-communicable disease affecting approximately 2-3% of the world's population, regardless of gender and age. In most cases (about 70-80%), the skin lesions are mild and do not require systemic treatment. The etiology of psoriasis development is not fully understood. In addition to genetic predisposition, the increased immune response in PS may be a consequence of systemic inflammation due to intestinal dysbiosis associated with increased intestinal permeability.

Dietary ingredients support skin health. Among them, prebiotics gained our special interest as ingredients with proven beneficial effects on host health by modulating gut microflora. Inulin-type fructans derived from chicory are prebiotics that favorably alters the composition and activity of the intestinal microbes and alleviates the inflammation in the intestines. The investigators supposed that restoring the balance of the gut microbiota and the proper functioning of the intestinal barrier in subjects with psoriasis will alleviate the inflammatory symptoms and skin lesions observed in this chronic dermatitis. The aim of the research is to determine whether dietary supplementation with inulin-type β-fructans derived from chicory will transfer health benefits to individuals with psoriasis and to investigate whether these benefits are due to modification of the composition or activity of the gut microbiota.

To achieve this goal, the original, advanced, and complex studies were proposed on subjects with psoriasis to investigate the effects of dietary inulin-type fructans on the characteristics of the gut microflora, metabolic parameters, and biomarkers of the skin-gut axis. The obtained results will provide new knowledge and explain the nature of the interaction between the gut microbiota and the skin, providing further clues about the functioning of the gut-skin axis.

ELIGIBILITY:
Inclusion Criteria for PS patients:

* mild psoriasis (PASI < 10),
* omnivorous diet,
* body mass index (BMI) 18 - 30 kg/m2
* general good health
* willing to give the written informed consent to participate the study

Exclusion Criteria for PS patients:

* other chronic or acute inflammatory skin diseases,
* gastrointestinal disease, cancer, cardiovascular complications, heart, kidney, and liver failure,
* bad or average overall health,
* positive tTG antibodies,
* currently receive anti-psoriatic systemic and biologic treatment,
* received antibiotics within previous month,
* use of dietary supplements containing probiotic, prebiotic, and/or symbiotic within previous month,
* Pregnancy, lactation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — women and men
Enrollment: 56 (Actual)
Dates: Start 2023-02-02 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Concentration of inflammatory mediators | 24 months
  The concentration of cytokines and chemokines: interferon-γ, interleukins: 1β, 1ra, 2, 4, 5, 6, 7, 8, 9, 10, 12 (p70), 13, 15, 17A, and tumor necrosis factor-α will be analyzed in blood using dedicated assay kit (Bio-Plex Pro Human Cytokine Assay; Bio-Rad)

SECONDARY OUTCOMES:
Assessment of the score of the psoriasis area and severity index (PASI) | 24 months
  The psoriasis area and severity index (PASI) combines the assessment of the severity of and area affected by psoriasis into a single score in the range 0 (no disease) to 72 (maximal disease).
Determination of the body mass index | 24 months
  The body height (in meters) and body weight (in kilograms) will be measeure and will be combined to report body mass index (BMI) in kg/m^2
Analysis of the concentration of anti-tissue transglutaminase antibodies | 24 months
  The concentration of anti-tissue transglutaminase antibodiesanty-tTG will be determined in blood serum according to standard procedures in the outpatient clinic of the Municipal Hospital in Olsztyn.
Analysis of the body composition | 24 months
  Body composition (percentage of total body fat, water, fat-free mass) will be assessed using a bioelectrical impedance analyser
Analysis of the concentration of C-reactive protein (CRP) | 24 months
  The concentration of the C-reactive protein (CRP) will be analyzed according to standard procedures in the outpatient clinic of the Municipal Hospital in Olsztyn. Serum anty-tTG will be determined to exclude the gluten-related disorders
Assessment of liver functions | 24 months
  The concentration of aspartate aminotransferase and alanine aminotransferase will be analyzed according to standard procedures in the outpatient clinic of the Municipal Hospital in Olsztyn.
Analysis of the concentration of creatinine | 24 months
  The concentration of creatinine will be analyzed in urine according to standard procedures in the outpatient clinic of the Municipal Hospital in Olsztyn.
Determination of carbohydrate metabolism | 24 months
  The concentration of glycated hemoglobin, glucose and insulin will be determined in fasting blood and analyzed according to standard procedures in the outpatient clinic of the Municipal Hospital in Olsztyn.
Determination of lipids metabolism | 24 months
  The concentration of apolipoproteins A and B will be determined in fasting blood and analyzed according to standard procedures in the outpatient clinic of the Municipal Hospital in Olsztyn.
Metabolic rate analysis | 24 months
  The resting energy expenditure will be measured by indirect respirometry with ventilated open-circuit (with canopy system) using Cosmed K5 mobile device, in conditions of thermal comfort, under fasting conditions, and in the supine position. Determining the volume of oxygen and carbon dioxide enables the determination of respiratory quotients and the degree of utilization of fat and carbohydrates in the body.
Assessment of qualitative and quantitative changes in the intestinal microbiota | 24 months
  The hyper-variable regions of the 16S rRNA bacterial gene (V3-V8) will be amplified. Bacterial libraries will be created using a Ligation Sequencing Kit 1D plus either Native Barcoding Expansion or a set of custom barcodes. Final libraries will be sequenced on a GridION X5 sequencer (Oxford Nanopore Technologies, Oxford, UK). High-quality reads will be processed for taxonomic identification by matching the NGS sequences with sequences deposited in the NCBI using a modified uSEARCH algorithm.
Assessment of the metabolic activity of intestinal microbiota | 24 months
  The concentration and profile of short-chain fatty acids (SCFA) will be analyzed using the gas chromatograph with a flame-ionization detector and the autosampler in stool samples collected from patients after nutritional intervention with prebiotic or placebo.
Determination of changes in the expression of genes of inflammatory response in skin | 24 months
  Changes in the expression of genes of inflammatory response will be determined by real-time PCR in skin biopsies collected from patients after nutritional intervention with prebiotic or placebo
Immunohistological skin analysis | 24 months
  The concentration of tumor necrosis factor-α, interleukins 17A, 17F, 12, 23, 8, 22, 35, and interferon-gamma will be determined in lesional and non-lesional skin specimens collected from study participants.
Determination of the concentration of biomarkers of intestinal barrier permeability and integrity | 24 months
  The concentration of the selected intestinal barrier permeability and integrity biomarkers will be analyzed using the ELISA method in the blood (zonulin, iFABP, claudin-3, bacterial LPS) and in stool (calprotectin, β-defensin-2, α1-Antitrypsin, sIgA) samples.
Determination of the activity of oxidative stress parameters | 24 months
  Superoxide dismutase activity and catalase activity will be analyzed in blood serum
Qualitative characteristics of volatile organic compounds | 24 months
  The profile of volatile organic compounds will be determined by headspace microextraction coupled with gas-chromatography and mass spectrometry in urine and stool samples
Determination of the nutritional status | 24 months
  Nutritional status will be evaluated based on Food Frequency Questionnaire and a 3-days food record

CONTACTS AND LOCATIONS:
Overall Officials: Urszula Krupa-Kozak, PhD, Principal Investigator — Institute of Animal Reproduction and Food Research of Polish Academy of Sciences in Olsztyn, Poland; Agnieszka Owczarczyk-Saczonek, Prof, Principal Investigator — Faculty of Medical Sciences of the University of Warmia and Mazury in Olsztyn, Poland; Ewa Lange, PhD, Principal Investigator — Institute of Human Nutrition Sciences, Warsaw University Of Life Sciences (SGGW), Poland
Locations (2):
- Poland (2):
  - Chair and Clinic of Dermatology, Sexually Transmitted Diseases and Clinical Immunology, Municipal Hospital Complex, al. Wojska Polskiego 30, Olsztyn
  - Institute of Animal Reproduction and Food Research, Polish Academy of Sciences, ul. Tuwima 10, Olsztyn

IPD SHARING:
Plan to Share IPD: No
Research results presented as average (+/- SD) or median will be successively made available in the form of English-language scientific publications in the Open Access format published in international journals and/or presented in the form of conference reports.